CLINICAL TRIAL: NCT06312449
Title: Effect of Peanut Balls Used on the Duration of the Second Stage of Labor, Pushing Perceptions, Fatigue and Birth Outcomes
Brief Title: Effect of Peanut Balls Used of the Second Stage of Labor, Pushing Perceptions, Fatigue and Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Yu-Ching (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Tung Yu-Ching, Linkou Chang Gung Memorial Hospital, Delivery Room, Vice Head Nurse, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2211110001
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Other
Keywords: Peanut ball; Second stage of labor; Perceived effort experience; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The experimental group (Experimental): The second stage of delivery involves using the lateral position with peanut ball
  Interventions: Other: The side-lying position with the peanut ball during the second stage of labor.
- Control Group A (Placebo Comparator): The second stage of delivery adopts the lateral position
  Interventions: Other: During the second stage, the patient is placed in a lateral position
- Control Group B (No Intervention): As usual care

INTERVENTIONS:
Other: The side-lying position with the peanut ball during the second stage of labor. — The usage of the peanut ball is divided into two stages:
  Stage one: The parturient assumes a side-lying position with the bed elevated to a 30-degree angle. The peanut ball is placed between the legs, allowing for leg separation. The parturient can choose to lie on either the left or right side according to preference.
  Stage two: When the fetal presenting part reaches 1 centimeter below the ischial spine (+1 Station), still in a side-lying position with the bed elevated to a 30-degree angle, the parturient has the option to switch sides. The peanut ball is then positioned between the legs with the knees bent together, for pushing
  Arms: The experimental group
Other: During the second stage, the patient is placed in a lateral position — The parturient assumes a side-lying position with the bed elevated to a 30-degree angle. The parturient can choose to lie on either the left or right side according to preference.When the fetal presenting part reaches 1 centimeter below the ischial spine (+1 Station), still in a side-lying position with the bed elevated to a 30-degree angle, the parturient has the option to switch sides, for pushing
  Arms: Control Group A

SUMMARY:
This study aims to explore the use of peanut balls during the second stage of labor. It compares three different positions: traditional lithotomy position, lateral position, and lateral position with peanut ball in terms of women's perceived pushing effort experiences, fatigue, and birth outcomes.

DETAILED DESCRIPTION:
The experimental research design involves enrolling participants during their hospitalization for childbirth. After explanation and consent, participants are sequentially assigned to Control Group B, Control Group A, and the Experimental Group. The Experimental Group receives education and guidance on using a peanut ball, while Control Groups receive standard care. During the second stage of labor, the Experimental Group assumes a side-lying position with the bed elevated at a 30-degree angle and uses the peanut ball with exertion. Control Group A assumes a side-lying position with the bed elevated at a 30-degree angle without the peanut ball, and Control Group B assumes a traditional lithotomy position with the bed elevated at a 30-degree angle with exertion.This study was conducted at a maternity ward in the Northern Region of a certain medical center. Participants were selected through consecutive convenient sampling.The total of 192 participants for the entire study.The research tools included:1.Personal basic demographic and obstetric information survey form: A self-designed questionnaire to gather personal basic information.2.Labor exertion experience scale: Adapted from the modified 10-item labor exertion experience scale designed by Chang et al. (2011).3.Visual Analog Scale for Fatigue (VAS-F): Employed as an assessment tool for fatigue.After enrollment, the experimental group received instructions on the intervention with the peanut ball. Research staff provided guidance using an educational leaflet on the purpose, timing, method, and precautions of using the peanut ball.Participants and their birth companions were required to demonstrate their understanding by performing the instructed actions, with corrections provided as necessary.

The research team members did not intervene during the execution process. Care was provided by instructed caregivers, who stayed with the parturients throughout the second stage of labor. Each group of participants was accommodated in individual labor rooms to prevent mutual interference. When the cervix was fully dilated to 10 centimeters or when the parturient felt a strong urge to push, or when the fetal presenting part reached 1 centimeter below the ischial spine (+1 Station), instruction on closed-glottis pushing for 5-6 seconds at a time began. The experimental group pushed in a side-lying position with the peanut ball, while Control Group A pushed in a side-lying position, and Control Group B pushed in a traditional lithotomy position. Within 1-4 hours postpartum, fatigue was assessed using the VAS-F at two time points (T1 and T2), and participants were instructed to complete the labor exertion experience scale. Finally, medical records and parturition records were transcribed to complete the labor duration and related data forms.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women with a singleton fetus in cephalic presentation at 36 weeks gestation or later.
* Anticipated vaginal delivery.
* Ability to understand, speak, read, and write Chinese.
* Normal prenatal examination findings for the fetus.
* Low-risk pregnancy.
* Voluntary participation after receiving an explanation of the study.

Exclusion Criteria:

* Mothers or fetuses experiencing abnormalities during labor requiring emergency cesarean section.
* Participants unwilling to engage in the side-lying position with exertion using the peanut ball during the second stage of labor.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
The duration of the second stage of labor of women who use side-lying with peanut balls. | calculated from the labor records within 24 hours postpartum, will be recorded by the researcher onto the individual basic information form.
  The duration of the second stage of labor
The pushing time of women in the second stage of labor who use side-lying with peanut balls. | As documented in the nursing records within 24 hours postpartum, will be transcribed by the researcher onto the second stage labor pushing record form.
  The second stage of labor pushing time
lateral position with peanut ball in terms of women's perceived pushing effort experiences. | Measurements will be conducted within 1 to 4 hours postpartum.
  Measuring pushing effort experiences
Parturients using the side-lying position with a peanut ball for experience levels of fatigue. | Measurements will be conducted within 1 to 4 hours postpartum.
  Measuring fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ching Tung, Nurse, Principal Investigator — Chang Gung Medical Foundation Institutional Review Board
Locations (1):
- Yu-Ching Tung, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No